CLINICAL TRIAL: NCT06693635
Title: Evaluating the Impact of Artificial Intelligence in Implant Planning Software: A Case Study Approach
Brief Title: Comparative Evaluation of Implant Planning Software
Status: Completed | Type: Observational
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, DDS, MSc, University of Bari Aldo Moro
Other Study IDs: AISoftware
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Edentulous Jaw; Edentulous Alveolar Ridge; Edentulous Mouth; Partial-edentulism
Keywords: Artificial Intelligence in Implantology; AI; Implant planning; AI software
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Implant planning — The implant planning will be carried out using various software programs. The AI assistance provided by each software will be evaluated.

SUMMARY:
Artificial intelligence (AI) is increasingly being integrated into dental implant planning, revolutionizing the way clinicians approach treatment. AI-driven software can enhance the accuracy of implant placement by analyzing complex data sets, including bone density, anatomical structures, and patient-specific factors. This technology enables the creation of precise 3D models and surgical guides, facilitating more predictable and personalized treatment outcomes. Additionally, AI algorithms can automate tasks such as segmentation, matching digital impressions with CBCT scans, and even suggesting optimal implant positions. The integration of AI in implant planning not only improves clinical efficiency but also contributes to better patient outcomes by reducing surgical risks and enhancing the overall success of implant procedures.

ELIGIBILITY:
Inclusion Criteria:

* CBCT of Patient who needs Implant rehabilitations

Exclusion Criteria:

* Patient not suitable for implant rehabilitation

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients requiring implant rehabilitation with digital planning
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Segmentation of Bones | 1 day
  The segmentation of bone structures and anatomical boundaries performed by the software will be evaluated.
Recognition of Neural structure | 1 day
  The segmentation and recognition of nerve structures performed by the software will be evaluated.
Segmentation of teeth | 1 day
  The segmentation of teeth performed by the software will be evaluated.
Bone density | 1 day
  The bone hardness and density data will be evaluated at three different points. The value will be given on the Hounsfield Scale.
Time Workflow | 1 day
  The execution time of each planning will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe D'Albis, Dr, Principal Investigator — University of Bari Aldo Moro; Massimo Corsalini, Prof, Study Director — University of Bari Aldo Moro; Saverio Capodiferro, Prof, Study Director — University of Bari Aldo Moro
Locations (1):
- University of Bari Aldo Moro, Bari, Italy